CLINICAL TRIAL: NCT01470833
Title: Non-operative Treatment of Acute Achilles Tendon Rupture Using Dynamic Rehabilitation. The Influence of Early Weight-bearing Compared With Non-weight-bearing
Brief Title: Non-operative Treatment of Acute Achilles Tendon Rupture Using Dynamic Rehabilitation. Influence of Early Weight-bearing Compared With Non-weight-bearing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Collaborators: DJO Incorporated (Industry)
Responsible Party: Principal Investigator, Kristoffer Barfod, Medical Doctor, Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ASR2011
Record Dates: First submitted 2011-11-09; First posted 2011-11-11 (Estimated); Last update posted 2013-08-20 (Estimated); Status verified 2013-08

CONDITIONS: Acute Achilles Tendon Rupture
Keywords: Achilles tendon; rupture; non-operative; treatment
MeSH Terms: conditions — Rupture

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Non-weight-bearing (No Intervention): The group of non-weightbearing is instructed as follows:
  Week 1 to 6 No weightbearing. Crutches are obligatory. Week 7 to 8 Full weightbearing is allowed.
  Dynamic rehabilitation From day 15 patients of both groups must do ankle exercises. Minimum 5 times a day the patient must take of the orthosis. Sitting at a table with the leg hanging freely over the edge a series of 25 active dorsal flexion and passive plantar flexion exercises must be made.
- Early weight-bearing (Experimental): The group allowed early weight-bearing is instructed as follows:
  Week 1 to 2 Weightbearing is allowed with in pain limit. Crutches are recommended.
  Week 3 to 4 Full weightbearing is allowed. Week 5 to 8 Full weightbearing is allowed. Crutches should be avoided.
  Interventions: Procedure: Early weight-bearing

INTERVENTIONS:
Procedure: Early weight-bearing — The group allowed early weight-bearing is instructed as follows:
  Week 1 to 2 Weight-bearing is allowed with in pain limit. Crutches are recommended.
  Week 3 to 4 Full weight-bearing is allowed. Week 5 to 8 Full weight-bearing is allowed. Crutches should be avoided.
  Dynamic rehabilitation From day 15 patients of both groups must do ankle exercises. Minimum 5 times a day the patient must take of the orthosis. Sitting at a table with the leg hanging freely over the edge a series of 25 active dorsal flexion and passive plantar flexion exercises must be made.
  Arms: Early weight-bearing

SUMMARY:
Acute achilles tendon rupture is relatively frequent (11 to 37 per 100,000). There are great social benefits in optimizing treatment and shortening recovery.

There is no consensus concerning the best treatment of acute achilles tendon rupture. Traditionally, surgical treatment is considered superior, but more recent studies show evidence that non-operative treatment with early dynamic rehabilitation gives the same functional outcome with fewer side effects.

Traditionally non-operative treatment involves non-weightbearing for 6 weeks. This is not evidence based rather due to tradition. It is well documented that mechanical load improves tendon healing in general and has no detrimental effect on the healing of operated achilles tendons.

The objective of this randomized study is to compare early weight-bearing with non-weight-bearing following non-operative treatment of acutely ruptured Achilles tendons.

DETAILED DESCRIPTION:
Background Acute achilles tendon rupture is relatively frequent (11 to 37 per 100,000) and potentially debilitating. Age distribution is bimodal, with a maximum incidence of sports-related injuries around 40 years of age. This is followed by a second and smaller increase in the incidence 50-60 years of age due to other, non sports-related injuries (1-3). The disease costs millions of dollars in treatment and lost earnings.

There is no consensus on the best treatment of acute achilles tendon rupture. It is the authors' belief that the decision on non-operative or operative treatment significantly differ between the orthopedic surgical departments and individual orthopedic surgeons.

Surgery is traditionally considered superior to conservative treatment due to a lower risk of rerupture of the achilles tendon (4). Despite the fact that surgery has a significantly increased risk of serious side effects such as deep infection (4). The decision of operative treatment is based on studies comparing surgical treatment and early dynamisation with non-operative treatment without dynamisation. Recent studies show increasing evidence that non-operative treatment with early dynamisation of the ankle gives the same functional outcome as operative treatment without significantly increased risk of rerupture (5.6). The same studies show that the overall complication rate is higher with surgery than with non-operative treatment. The surgical complications include infection, nerve damage, adhesion, contracture and cosmetic problems.

Pajala et. al have compared outcome for patients who suffered rerupture with those who suffered a deep wound infection. They conclude that outcome after rerupture without complicating infection is satisfactory, whereas the outcome after deep wound infection is devastating (7). The risk of a debilitating complication is thus greater with surgery than is the case for conservative treatment.

Traditionally non-operative treatment involves non-weightbearing for 6 weeks. This is not evidence based rather due to tradition. Suchak et. al have shown that early weight bearing after surgical treatment of ASR improves health related quality of life in the period after surgery and has no negative effect on tendon healing.(9) It is well documented that mechanical load improves tendon healing (10). Thus it is reasonable to believe that early loading of the tendon under controlled conditions will affect tendon healing beneficially.

Objective of the study Primary purpose The objective of this randomized study is to compare early weight-bearing with non-weight-bearing following non-operative treatment of acutely ruptured Achilles tendons.

All patients are treated with dynamic rehabilitation in a DJO Walker orthosis. Functional outcome is self assessed using Achilles tendon Total Rupture Score (ATRS) and biomechanically by quantification of the stiffness of the achilles tendon and force development at concentric and eccentric work.

Secondary objectives Rerupture, time to return to work, time to return to sports.

Method and subjects:

The survey is conducted as a clinical randomized trial (RCT). Patients allowed to bear weight from day 1 are compared with patients who are not allowed to bear weight the first 6 weeks of treatment. The orthosis is equipped with a pressure sensor that detects when the patient bear weight on the foot. The project has been approved by the medical ethic committee.

Population 30 persons will be included in each group. Altogether 60 persons will be included.

Timeplan The study is planned for a period of 3 years. Recruitment of patients started 1st of April 2011 and is expected to be completed in 2012. The follow up period is 2 years.

Procedures In the emergency room an ankle orthosis (DJO Walker) is applied with the foot in 30 degree plantar flexion. The orthosis is worn for 8 weeks gradually bringing the foot to 0 degrees. From day 15 dynamisation of the ankle joint is performed.

Treatment Week 1 to 2 3 wedges. The orthosis must be worn 24 hours a day. Can not be removed by bathing or at night.

Week 3 to 4 2 wedges. Dynamic rehabilitation. The boot can not be removed at night.

Week 5 to 6 1 wedge. Dynamic rehabilitation. The boot can not be removed at night.

Week 7 to 8 No wedges. Dynamic rehabilitation. The boot can be removed at night.

The group allowed early weight-bearing is instructed as follows:

Week 1 to 2 Weightbearing is allowed with in pain limit. Crutches are recommended.

Week 3 to 4 Full weightbearing is allowed. Week 5 to 8 Full weightbearing is allowed. Crutches should be avoided.

The group of non-weightbearing is instructed as follows:

Week 1 to 6 No weightbearing. Crutches are obligatory. Week 7 to 8 Full weightbearing is allowed.

Dynamic rehabilitation From day 15 patients of both groups must do ankle exercises. Minimum 5 times a day the patient must take of the orthosis. Sitting at a table with the leg hanging freely over the edge a series of 25 active dorsal flexion and passive plantar flexion exercises must be made.

Verification of compliance All DJO walkers used in the study are equipped with an integrated pressure sensor that detects when load is applied in the boot.

Rehabilitation After 8 weeks the patient is seen at the out patient clinic. They are instructed rehabilitation regime by a physiotherapist. Rehabilitation is designed as a home exercise program with emphasis on movement, stability, coordination and strength.

Week 9 to 16 The patient may cycle and swim. Week 16 to 26 Jogging on soft surfaces. Week 26 Sports can be resumed. We do not recommend badminton, tennis and squash as well as contact sports before week 40 - 52. Week 52 No restrictions

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years.
* The patient must be able to speak and understand Danish.
* The patient must be able to give informed consent.
* The patient should be able to follow a regimen with a removable ankle orthosis.
* The patient must be able to determine when rupture occurred, and it can't be over 4 days old.
* The patient should be able to follow the postoperative controls.

Exclusion Criteria:

* Terminal illness.
* Former achilles tendon rupture
* Former surgery on the achilles tendon
* Treatment with fluoroquinolones during the last 6 months.
* Tendinosis treated with a tablet or injection with corticosteroids within the last 6 months.
* Diagnosis of arterial insufficient in the leg.
* Lack of palpable pulse in the foot
* Severe medical illness: ASA score greater than 2
* Distance from calcaneus to the rupture is less than 1 cm

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2011-04; Primary Completion 2013-04 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
ATRS (Achilles Tendon Total Rupture Score) | 1 year
  Patient-reported validated scoring tool developed for assessment of symptoms and physical activity after treatment for acute achilles tendon rupture.

SECONDARY OUTCOMES:
Heel-rise-work test | 1 year
  The accummulated work made doing repetetive heel-rises is messured on each leg.

CONTACTS AND LOCATIONS:
Overall Officials: Kristoffer W Barfod, Medical Doctor, Study Chair — Hvidovre University Hospital
Locations (1):
- Hvidovre Hospital, Copenhagen, Denmark